CLINICAL TRIAL: NCT00088881
Title: A Phase II Trial of R-CHOP Followed by Zevalin Radioimmunotherapy for Patients With Previously Untreated Stages I and II CD20+ Diffuse Large Cell Non-Hodgkin's Lymphoma
Brief Title: Rituximab, Combination Chemotherapy, and 90-Yttrium Ibritumomab Tiuxetan for Patients With Stage I or II Non-Hodgkin's Lymphoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02957; E3402 (Other: Eastern Cooperative Oncology Group (ECOG)); U10CA021115 (NIH)
Record Dates: First submitted 2004-08-04; First posted 2004-08-05 (Estimated); Results first posted 2015-02-18 (Estimated); Last update posted 2017-05-25 (Actual); Status verified 2017-04

CONDITIONS: Contiguous Stage II Adult Diffuse Large Cell Lymphoma; Extranodal Marginal Zone B-cell Lymphoma of Mucosa-associated Lymphoid Tissue; Nodal Marginal Zone B-cell Lymphoma; Noncontiguous Stage II Adult Diffuse Large Cell Lymphoma; Splenic Marginal Zone Lymphoma; Stage I Adult Diffuse Large Cell Lymphoma; Testicular Lymphoma; Waldenström Macroglobulinemia
MeSH Terms: conditions — Lymphoma, B-Cell, Marginal Zone; Lymphoma, Large B-Cell, Diffuse; Waldenstrom Macroglobulinemia | interventions — Rituximab; Prednisone; Cyclophosphamide; Doxorubicin; Vincristine; Indium; Radiotherapy; Radiation; Magnetic Resonance Spectroscopy; 2-phenyl-6-(2'-(4'-(ethoxycarbonyl)thiazolyl))thiazolo(3,2-b)(1,2,4)triazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (Experimental): R-CHOP (Rituximab, Cyclophosphamide, Doxorubicin, Vincristine, Prednisone): Patients receive R-CHOP every 21 days for 2 courses in the absence of disease progression or unacceptable toxicity. Patients achieving a complete response after 2 courses receive 2 additional courses. Patients achieving a partial response, uncertain CR, or stable disease receive 4 additional courses. Patients with progressive disease go off study.
  Zevalin™Radioimmunotherapy: Beginning no more than 9 weeks after the last course of R-CHOP, patients receive rituximab IV on day 1 followed by indium In 111 ibritumomab tiuxetan IV over 10 minutes for imaging studies. Patients then receive rituximab IV followed by yttrium Y 90 ibritumomab tiuxetan IV over 10 minutes on day 8.
  Radiation therapy: Patients with residual disease by CT scan or positron emission tomography (PET) scan after 12 weeks after radioimmunotherapy undergo conventional involved-field radiotherapy.
  Interventions: Biological: rituximab; Drug: prednisone; Drug: cyclophosphamide; Drug: doxorubicin; Drug: vincristine; Radiation: indium In 111 ibritumomab tiuxetan; Radiation: radiation therapy; Procedure: positron emission tomography

INTERVENTIONS:
Biological: rituximab — Given IV
  Other Names: IDEC-C2B8; IDEC-C2B8 monoclonal antibody; Mabthera; MOAB IDEC-C2B8; Rituxan
Drug: prednisone — Given orally
  Other Names: DeCortin; Deltra
Drug: cyclophosphamide — Given IV
  Other Names: CPM; CTX; Cytoxan; Endoxan; Endoxana
Drug: doxorubicin — Given IV
  Other Names: ADM; ADR; Adria; Adriamycin PFS; Adriamycin RDF
Drug: vincristine — Given IV
  Other Names: leurocristine sulfate; VCR; Vincasar PFS
Radiation: indium In 111 ibritumomab tiuxetan — Given IV
  Other Names: IDEC-In2B8
Radiation: radiation therapy — Undergo radiotherapy
  Other Names: irradiation; radiotherapy; therapy, radiation
Procedure: positron emission tomography — Undergo PET scans
  Other Names: FDG-PET; PET; PET scan; tomography, emission computed

SUMMARY:
This phase II trial is studying how well giving rituximab together with combination chemotherapy and 90-Yttrium ibritumomab tiuxetan works in treating patients with stage I or stage II lymphoma. Drugs used in chemotherapy, such as prednisone, cyclophosphamide, doxorubicin, and vincristine, work in different ways to stop cancer cells from dividing so they stop growing or die. Monoclonal antibodies such as rituximab and yttrium 90-Yttrium ibritumomab tiuxetan can locate cancer cells and either kill them or deliver radioactive cancer-killing substances to them without harming normal cells. Combining a monoclonal antibody with combination chemotherapy and a radiolabeled monoclonal antibody may kill more cancer cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the complete response rate (CR) and functional CR rate in patients with previously untreated stage I (with at least 1 risk factor) or stage II CD20+ diffuse large cell lymphoma who receive therapy with R-CHOP followed by 90-Yttrium -Zevalin™.

SECONDARY OBJECTIVES:

I. To evaluate the time to treatment failure, duration of response, and overall survival in these patients who receive therapy with R-CHOP followed by 90-Yttrium -Zevalin™.

II. To evaluate the toxicity of this therapy. III. To evaluate the toxicity of adding involved field radiation therapy > 12 weeks after Zevalin™ for patients with CT+/PET+ residual masses.

TERTIARY OBJECTIVES:

I. To evaluate PET scans pre -and post - R-CHOP/Zevalin™ therapy.

OUTLINE:

R-CHOP (rituximab, prednisone, cyclophosphamide, doxorubicin,vincristine): Patients receive oral prednisone once daily on days 1-5. Patients also receive rituximab IV over several hours followed by cyclophosphamide IV, doxorubicin IV, and vincristine IV over 30-60 minutes on day 1. Treatment repeats every 21 days for 2 courses in the absence of disease progression or unacceptable toxicity. Patients achieving a complete response (CR) after 2 courses receive 2 additional courses. Patients achieving a partial response, uncertain CR, or stable disease receive 4 additional courses. Patients are evaluated 3 weeks after the last course of therapy. Patients with progressive disease go off study.

Radioimmunotherapy: Beginning no more than 9 weeks after the reevaluation (or 12 weeks after the last dose of R-CHOP), patients receive rituximab IV on day 1 followed by indium In 111 ibritumomab tiuxetan IV over 10 minutes for imaging studies. Patients then receive rituximab IV followed by yttrium 90-Yttrium ibritumomab tiuxetan IV over 10 minutes on day 8.

Radiotherapy: Patients with residual disease by CT scan or positron emission tomography (PET) scan after 12 weeks after radioimmunotherapy undergo conventional involved-field radiotherapy.

Patients are followed every 3 months for 1 year, every 4 months for 1 year, every 6 months for 3 years, and then annually for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed diagnosis of diffuse large cell lymphoma
* Patients must be stage I or II (Modified Ann Arbor staging)
* Baseline measurements and evaluations must be obtained within 4 weeks of registration to the study; abnormal PET scans will not constitute evaluable disease unless verified by CT scan or other appropriate imaging; patients must have at least one objective measurable disease parameter (a lesion with at least 1 dimension > 1.5 cm); or if they are stage 1
* Stage I patients must have at least one of the following risk factors:

  * Age >= 60 years
  * Bulky disease (>= 5 cm in at least one dimension)
  * Elevated Lactate Dehydrogenase (LDH) above institutional upper limit of normal
  * Eastern Cooperative Oncology Group (ECOG) performance status = 2
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Absolute neutrophil count >= 1500/mm^3 (includes neutrophils and bands)
* Platelet count >= 100,000/mm^3
* Creatinine < 2.0 mg/dl
* Total bilirubin < 2 mg/dl (may be up to 3.0 mg/dl if due to liver involvement by lymphoma); patients with elevated total bilirubin should have a direct bilirubin checked; if the direct bilirubin is normal there is no need for a dose reduction
* Patients must have left ventricular ejection fraction (LVEF) of > 45%
* Patients must be tested for hepatitis B (HBV) surface antigen within 2 weeks of registration

  * NOTE: Patients who test positive will be allowed to participate but must be followed closely for clinical and laboratory signs of active HBV infection and for signs of hepatitis

Exclusion Criteria:

* Prior chemotherapy, radiation therapy, radioimmunotherapy, or immunotherapy; a short course (=< 14 days prior to registration) of corticosteroids is allowed
* Evidence of other malignancy:

  * Prior chemotherapy or prior radiation therapy for other malignancies
  * Currently receiving hormone therapy or chemotherapy for another malignancy even if the treatment is being provided in the adjuvant treatment setting, i.e. with no evidence of the original other malignancy
  * Adjuvant hormonal therapy must have been discontinued > 3 months before entering this study
  * Patients are eligible if they meet the following conditions: (a) treated carcinoma-in-situ of the cervix; (b) treated squamous cell or basal cell skin cancer; or (c) any other surgically cured malignancy from which the patient has been disease free for at least 3 years
* Pregnant or breast feeding, as there would be radiation exposure to the fetus or child; a negative pregnancy test is required =< 1 week prior to registration for women of childbearing potential (WOCBP). Women of childbearing potential and sexually active males must be strongly advised to use an accepted and effective method of contraception
* Known central nervous system (CNS) lymphoma, testicular lymphoma, or vitreous lymphoma
* Known HIV infection. The safety of Zevalin™ in this population has not been tested at this time
* Serious coexisting medical condition or active infection which would compromise the ability to deliver standard R-CHOP chemotherapy
* Evidence of myelodysplasia on bone marrow aspiration and biopsy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2004-12; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Witzig, Principal Investigator — Eastern Cooperative Oncology Group
Locations (1):
- Eastern Cooperative Oncology Group, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment: R-CHOP: Patients receive R-CHOP every 21 days for 2 courses in the absence of disease progression or unacceptable toxicity. Patients achieving a complete response (CR) after 2 courses receive 2 additional courses. Patients achieving a partial response, uncertain CR, or stable disease receive 4 additional courses. Patients are evaluated 3 weeks after the last course of therapy. Patients with progressive disease go off study.
  Zevalin™Radioimmunotherapy: Beginning no more than 9 weeks after the last course of R-CHOP, patients receive rituximab IV on day 1 followed by indium In 111 ibritumomab tiuxetan IV over 10 minutes for imaging studies. Patients then receive rituximab IV followed by yttrium Y 90 ibritumomab tiuxetan IV over 10 minutes on day 8.
  Radiotherapy: Patients with residual disease by CT scan or positron emission tomography (PET) scan after 12 weeks after radioimmunotherapy undergo conventional involved-field radiotherapy.
Period: Step 1 - R-CHOP
Arm/Group | Treatment
Started | 62
Eligible and Treated | 53
Completed | 48
Not Completed | 14
Not completed — Patient ineligible | 9
Not completed — Adverse Event | 1
Not completed — Withdrawal by Subject | 2
Not completed — Physician Decision | 1
Not completed — Insurance company refused to cover | 1
Period: Step 2 - Zevalin™ Radioimmunotherapy
Arm/Group | Treatment
Started | 56 (This includes all patients who received step 2 treatment regardless of eligibility.)
Eligible and Treated | 48
Completed | 45
Not Completed | 11
Not completed — Patient ineligible | 8
Not completed — Other | 3
Period: Step 3 - Radiation Therapy
Arm/Group | Treatment
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Eligible and treated patients
Arm/Group | Treatment
Number analyzed (Participants) | 53
Age, Continuous [Median (Full Range); unit: years] | 62 [20 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 32

OUTCOME MEASURES:

1. Primary Outcome: Complete Response (CR) +Complete Response/Uncertain (CRu) in Patients Treated With R-CHOP Followed by 90-Yttrium -Zevalin™.
Description: Response was assessed based upon the criteria from the International Workshop to Standardize Criteria for Non-Hodgkin's Lymphoma (Cheson, 1999). CR is defined as complete disappearance of all detectable clinical and radiographic evidence of disease and disappearance of all disease related B-symptoms if present prior to therapy, as well as normalization (normal limits of institutional labs) of those biochemical abnormalities (e.g., LDH) definitely attributed to NHL. CRu is defined as meeting the criteria of CR except one or more of the followings: A residual dominant node (or extra-nodal mass) that is currently > 1.5 cm in greatest diameter that has decreased by > 75% from baseline in the product of its diameters. Individual dominant nodes (or extra-nodal masses) that were previously confluent must have decreased by > 75% in SPD compared with the size of the original mass. Indeterminate bone marrow (increased number or size of aggregates without cytologic or architectural atypia).
Time Frame: Assessed after 2 cycles of R-CHOP, after completion of R-CHOP, and at Week 12 After 90-Yttrium Zevalin
Population: Eligible and treated patients
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Treatment
Number analyzed (Participants) | 53
proportion of participants | 0.87 [0.75 to 0.95]

2. Primary Outcome: Functional CR in Patients Treated With R-CHOP Followed by 90-Yttrium -Zevalin™.
Description: Patients will be considered a functional CR if they meet the criteria for a CR, or if they meet the criteria for a CRu or partial response (PR) by CT and are PET negative. Please see primary outcome #1 for the definition of CR and CRu. PR is defined as: A decrease of >50% in the SPD (sum of products of the diameters) of the six largest (or less) dominant nodes or extra-nodal masses. No increase in the size of the liver or the spleen. No unequivocal progression in any non-measurable or non-dominant site. Splenic and hepatic nodules must regress by >50% in SPD (sum of the products of the diameters). Bone marrow assessment is not relevant for determination of a PR because it is assessable and not measurable disease. No new sites of disease.
Time Frame: Assessed after 2 cycles of R-CHOP, after completion of R-CHOP, and at Week 12 After 90-Yttrium Zevalin
Population: Eligible and treated patients.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Treatment
Number analyzed (Participants) | 53
proportion of participants | 0.89 [0.77 to 0.96]

3. Secondary Outcome: 3-year Time to Treatment Failure (TTF) Rate
Description: Time to treatment failure (TTF) is defined as the time from step 1 registration to disease progression or death. TTF is censored at last documented progression free for cases without progression. The 3-year TTF rate is defined as the probability of patients remaining free from treatment failure at 3 years.
Time Frame: Assessed every 3 months for one year; every 4 months for the second year; then every 6 months for 3 years; then annually to 10 years from patient entry.
Population: Eligible and treated patients
Measure: Number (95% Confidence Interval); unit: probability
Arm/Group | Treatment
Number analyzed (Participants) | 53
probability | 0.92 [0.84 to 1.00]

4. Secondary Outcome: 3-year Overall Survival (OS) Rate
Description: Overall survival (OS) is defined as the time from step 1 registration to death of any cause. OS is censored at the date last known alive for cases that are alive. The 3-year OS rate is defined as the probability of patients remaining alive at 3 years.
Time Frame: Assessed every 3 months for 2 years, then every 6 months for 3 years; then annually to 10 years from patient entry.
Population: Eligible and treated patients
Measure: Number (95% Confidence Interval); unit: probability
Arm/Group | Treatment
Number analyzed (Participants) | 53
probability | 0.98 [0.94 to 1.00]

ADVERSE EVENTS:
Time Frame: Assessed every 3 weeks while on treatment and for 30 days after the end of treatment
Groups:
- Step 1 - R-CHOP: Patients receive R-CHOP every 21 days for 2 courses in the absence of disease progression or unacceptable toxicity. Patients achieving a complete response (CR) after 2 courses receive 2 additional courses. Patients achieving a partial response, uncertain CR, or stable disease receive 4 additional courses. Patients are evaluated 3 weeks after the last course of therapy. Patients with progressive disease go off study.
- Step 2 - Zevalin™ Radioimmunotherapy: Beginning no more than 9 weeks after the last course of R-CHOP, patients receive rituximab IV on day 1 followed by indium In 111 ibritumomab tiuxetan IV over 10 minutes for imaging studies. Patients then receive rituximab IV followed by yttrium Y 90 ibritumomab tiuxetan IV over 10 minutes on day 8.
- Step 3 - Radiation Therapy: Patients with residual disease by CT scan or positron emission tomography (PET) scan after 12 weeks after radioimmunotherapy undergo conventional involved-field radiotherapy.
Arm/Group | Step 1 - R-CHOP | Step 2 - Zevalin™ Radioimmunotherapy | Step 3 - Radiation Therapy
Serious Adverse Events (participants affected / at risk) | 44/62 | 46/56 | 0/1
Other Adverse Events (participants affected / at risk) | 62/62 | 55/56 | 0/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Step 1 - R-CHOP (N=62) | Step 2 - Zevalin™ Radioimmunotherapy (N=56) | Step 3 - Radiation Therapy (N=1)
Allergic reaction (Immune system disorders) | 1 | 0 | 0
CD4 decreased (Investigations) | 0 | 1 | 0
Anemia (Blood and lymphatic system disorders) | 5 | 3 | 0
Leukocytes decreased (Investigations) | 22 | 20 | 0
Lymphopenia (Investigations) | 26 | 34 | 0
Neutrophils decreased (Investigations) | 27 | 29 | 0
Platelets decreased (Investigations) | 5 | 26 | 0
Heart block Stokes-Adams syndrome (Cardiac disorders) | 0 | 0 | 0
Hypotension (Vascular disorders) | 1 | 0 | 0
Fatigue (General disorders) | 7 | 0 | 0
Nail changes (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Anorexia (Metabolism and nutrition disorders) | 4 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 1 | 0
Diarrhea w/o prior colostomy (Gastrointestinal disorders) | 1 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0
Muco/stomatitis by exam, oral cavity (Gastrointestinal disorders) | 1 | 0 | 0
Muco/stomatitis (symptom) oral cavity (Gastrointestinal disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 10 | 0 | 0
Infection w/ gr3-4 neut, lung (Infections and infestations) | 2 | 0 | 0
Infection w/ gr3-4 neut, skin (Infections and infestations) | 0 | 1 | 0
Infection w/ gr3-4 neut, blood (Infections and infestations) | 1 | 0 | 0
Acidosis (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypocalcemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Creatinine increased (Investigations) | 1 | 0 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 6 | 0 | 0
Hypoglycemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypomagnesemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypophosphatemia (Metabolism and nutrition disorders) | 2 | 0 | 0
Hypokalemia (Metabolism and nutrition disorders) | 2 | 0 | 0
Hyponatremia (Metabolism and nutrition disorders) | 1 | 0 | 0
Nonneuropathic generalized weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Neuropathy-sensory (Nervous system disorders) | 3 | 1 | 0
Psychosis (Psychiatric disorders) | 2 | 0 | 0
Syncope (Nervous system disorders) | 3 | 0 | 0
Bladder, pain (Renal and urinary disorders) | 1 | 0 | 0
Face, pain (General disorders) | 1 | 0 | 0
Neuropathic, pain (Nervous system disorders) | 0 | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Pulmonary/Upper Respiratory-other (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Step 1 - R-CHOP (N=62) | Step 2 - Zevalin™ Radioimmunotherapy (N=56) | Step 3 - Radiation Therapy (N=1)
Anemia (Blood and lymphatic system disorders) | 48 | 44 | 0
Leukocytes decreased (Investigations) | 39 | 51 | 0
Lymphopenia (Investigations) | 50 | 47 | 0
Neutrophils decreased (Investigations) | 28 | 41 | 0
Platelets decreased (Investigations) | 20 | 51 | 0
Fatigue (General disorders) | 50 | 32 | 0
Fever w/o neutropenia (General disorders) | 0 | 3 | 0
Insomnia (Psychiatric disorders) | 6 | 0 | 0
Rigors/chills (General disorders) | 7 | 0 | 0
Sweating (Skin and subcutaneous tissue disorders) | 5 | 0 | 0
Weight loss (Investigations) | 11 | 3 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 31 | 7 | 0
Pruritus/itching (Skin and subcutaneous tissue disorders) | 6 | 0 | 0
Rash/desquamation (Skin and subcutaneous tissue disorders) | 11 | 0 | 0
Anorexia (Metabolism and nutrition disorders) | 14 | 4 | 0
Constipation (Gastrointestinal disorders) | 35 | 0 | 0
Diarrhea w/o prior colostomy (Gastrointestinal disorders) | 16 | 6 | 0
Dry mouth (Gastrointestinal disorders) | 6 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 19 | 0 | 0
Muco/stomatitis by exam, oral cavity (Gastrointestinal disorders) | 14 | 0 | 0
Muco/stomatitis (symptom) oral cavity (Gastrointestinal disorders) | 17 | 0 | 0
Nausea (Gastrointestinal disorders) | 37 | 6 | 0
Taste disturbance (Nervous system disorders) | 12 | 3 | 0
Vomiting (Gastrointestinal disorders) | 15 | 0 | 0
Edema limb (General disorders) | 6 | 0 | 0
Alkaline phosphatase increased (Investigations) | 13 | 8 | 0
Alanine aminotransferase increased (Investigations) | 4 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 9 | 4 | 0
Blood bilirubin increased (Investigations) | 0 | 3 | 0
Hypocalcemia (Metabolism and nutrition disorders) | 5 | 0 | 0
Creatinine increased (Investigations) | 4 | 0 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 44 | 16 | 0
Hypokalemia (Metabolism and nutrition disorders) | 4 | 0 | 0
Dizziness (Nervous system disorders) | 7 | 0 | 0
Neuropathy-motor (Nervous system disorders) | 6 | 0 | 0
Neuropathy-sensory (Nervous system disorders) | 38 | 10 | 0
Abdomen, pain (Gastrointestinal disorders) | 6 | 0 | 0
Head/headache (Nervous system disorders) | 8 | 3 | 0
Joint, pain (Musculoskeletal and connective tissue disorders) | 4 | 0 | 0
Muscle, pain (Musculoskeletal and connective tissue disorders) | 9 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 7 | 0 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 8 | 4 | 0
Voice changes/dysarthria (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less